CLINICAL TRIAL: NCT00979173
Title: A Pharmacokinetic Study of AC480 Administered Twice Daily in Surgically Resectable Malignant Glioma Patients Not on Enzyme-Inducing Anticonvulsants
Brief Title: Pharmacokinetics (PK) Study of AC480 for Recurrent Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Annick Desjardins (Other)
Collaborators: Ambit Biosciences Corporation (Industry)
Responsible Party: Sponsor-Investigator, Annick Desjardins, Assist Professor of Medicine-Neurology, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00018751
Record Dates: First submitted 2009-08-06; First posted 2009-09-17 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2013-12

CONDITIONS: Glioma
Keywords: malignant glioma; glioblastoma multiforme; gliosarcoma; anaplastic astrocytoma; anaplastic oligodendroglioma; anaplastic mixed glioma; Pro00018751; Duke; Ambit; AC480
MeSH Terms: conditions — Glioma; Glioblastoma; Gliosarcoma; Astrocytoma; Oligodendroglioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AC480 (Experimental): Patients who are not on enzyme inducing anti-epileptic drugs (EIAEDs) and are scheduled to undergo salvage surgical resection treated with preoperative AC480 at 300 mg BID followed by post-surgical AC480 at 300 mg BID.
  Interventions: Drug: AC480

INTERVENTIONS:
Drug: AC480 — Subjects will be initiated on AC480 300mg orally BID for 14 (+/-2 days) before surgery. After surgery, subjects will continue to be dosed with AC480 until either disease progression or intolerance, and will be evaluated every other cycle (i.e., every 4 weeks).

SUMMARY:
The primary objective is to evaluate the intratumoral and plasma pharmacokinetics of AC480 among patients who are candidates for a resection with a recurrent malignant glioma who are not on CYP-3A enzyme inducing anti-epileptic drugs (EIAEDS). Secondary objectives include the following: to evaluate the antiproliferative effect of AC480 by FDG-PET Scan; to evaluate the safety and tolerability of AC480; and, to describe 6-month progression-free survival (PFS) and radiographic response.

This is a single institution, open label, pharmacokinetic study of AC480 in patients with recurrent malignant glioma. The study will enroll 5 patients who are not on enzyme inducing anti-epileptic drugs (EIAEDs) and are scheduled to undergo salvage surgical resection for preoperative treatment with AC480 at 300 mg orally twice daily (BID) for 14 (plus or minus 2) days before surgery (Part I- Induction Therapy). After surgery (Part II- Maintenance Therapy), patients will continue to be dosed with AC480 until disease progression or intolerance, and will be evaluated after every other cycle (1 cycle is 28 days).

DETAILED DESCRIPTION:
Plasma and tumoral pharmacokinetics, as well as FDG-PET data will be analyzed to determine the intratumoral and plasma levels of AC480 obtained and its antiproliferative activity. After recovery from surgery, all patients will resume AC480 at 300 mg orally BID until evidence of disease progression or toxicity (Part II: Maintenance Therapy). Those patients will be followed for determination of 6-month progression free survival. Patients will remain on treatment for as long as they have clinical benefit from the treatment. There will be no limit to the number of cycles of treatment a patient can receive providing they continue to benefit from and are not intolerant to AC480 administration.

The data collected in this study will be summarized in tables listing the mean, standard deviation, and number of patients for continuous data, or in tables listing count and percentage for categorical data, where appropriate. All patient data will be listed by patient or by parameter, all statistical analyses will be performed and all data appendices will be created by using the SAS system. Pharmacokinetic analysis will be made to determine if AC480 reaches the intracerebral tumor tissue. Comparisons will be made between the data obtained from the plasma of the same patients treated on AC480, including determination of the tumor-to-plasma ratio. The most common side effects of AC480 are generally mild to moderate in severity and include: nausea, vomiting, diarrhea, fatigue, cough, elevation of the liver enzymes, anemia, and rash.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of a recurrent/progressive WHO grade 4 malignant glioma (glioblastoma multiforme or gliosarcoma) or WHO grade 3 malignant glioma (anaplastic astrocytoma, anaplastic oligodendroglioma or anaplastic mixed glioma) and be surgical candidates. Recurrence will be defined based on the modified MacDonald criteria or based on histopathologic confirmation of tissue obtained via surgical intervention. Patients with prior low-grade glioma are eligible if histologic assessment demonstrates transformation to WHO grade III or IV malignant glioma.
* Greater than or equal to 18 years old.
* Karnofsky Performance Status (KPS) greater than or equal to 60%.
* Patients must be presenting in first, second or third relapse. Relapse is defined as progression following anti-cancer therapy other than surgery, including non-surgical therapies that are considered standard treatment for high-grade glioma if administered to patients with prior low-grade glioma. Prior therapy must have included external beam radiotherapy.
* Adequate bone marrow, liver and renal function as assessed by the following:

  * Hematocrit > or = to 29%
  * Absolute neutrophil count (ANC) > or = to 1,500/mL
  * Platelet count > or = to 125,000/mL
  * Total bilirubin < or = to 1.5 x ULN
  * ALT and AST < or equal to 2.5 x the ULN
  * INR < 1.5 or a PT/PTT within normal limits (unless on therapeutic anti-coagulation). Patients receiving anti-coagulation treatment with a low-molecular weight heparin will be allowed to participate, however oral warfarin is not permitted except for low-dose warfarin (1mg po DAILY).
  * Creatinine < or = to 1.5 x ULN
  * Serum Na, K+, Mg2+, Phosphate and Ca2+ Within Normal Limit (WNL)
* An interval of at least 12 weeks from completion of standard, daily XRT, unless one of the following occurs: a) new area of enhancement on MRI imaging that is outside the XRT field; b) biopsy proven recurrent tumor; c) radiographic evidence of progressive tumor on 2 consecutive scans at least 4 weeks apart.
* An interval of at least 4 weeks from prior chemotherapy (except nitrosoureas which require 6 weeks) unless there is unequivocal evidence of tumor progression and the patient has recovered from all anticipated toxicities from prior therapy.
* An interval of a least 4 weeks from exposure to investigational agents, unless there is unequivocal evidence of tumor progression and the patients has recovered from all anticipated toxicities from prior therapy.
* Signed written informed consent including HIPAA language according to institutional guidelines. This informed consent shall include language whereby Ambit shall have access to the patient's protected health information. A signed informed consent must be obtained prior to any study specific procedures.
* If sexually active, patients will take contraceptive measures for the duration of the treatments and for 3 months following discontinuation of AC480.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (sensitivity < or = to 25IU HCG/L) within 72 hours prior to the start of study drug administration. Males and females age ≥ 18 years. WOCBP include any female that has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not post menopausal (defined as amenorrhea > 12 consecutive months; or women on hormone replacement therapy [HRT] with documented serum follicle stimulating hormone [FSH] level > 35 mIU/mL). Even women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or are practicing abstinence or where the partner is sterile (e.g., vasectomy), should be considered to be of childbearing potential.
* Patients having received bevacizumab are eligible four weeks after the last dose of bevacizumab.

Exclusion Criteria:

* Subjects on enzyme-inducing antiepileptic drugs (phenytoin, phenobarbitol, carbamazepine, oxcarbamazepine, and primidone).
* Subjects previously treated with targeted therapies to EGFR and HER2.
* More than 3 prior episodes of progressive disease.
* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 3 months after completion of the study.
* Women who are pregnant or breastfeeding.
* Men who are unwilling or unable to use an acceptable method of birth control if their sexual partners are WOCBP for the entire study period and for at least 3 months after completion of the study.
* A serious uncontrolled medical disorder or active infection requiring IV antibiotics, which would impair the ability of the subject to receive protocol therapy.
* Uncontrolled or significant cardiovascular disease, including:

  * A myocardial infarction within 12 months;
  * Uncontrolled angina within 6 months;
  * Congestive heart failure NYHA class 3 or 4, or subjects with history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram (ECHO) performed within 3 months prior to study entry results in a left ventricular ejection fraction (LVEF) that is ≥ 45%;
  * Diagnosed or suspected long QT syndrome;
  * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes);
  * Any subject with a history of any arrhythmia should be discussed with the Ambit Medical Monitor prior to entry into the study;
  * Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec);
  * Any history of second or third degree heart block;
  * Heart rate < 50 / minute on pre-entry electrocardiogram;
  * Uncontrolled hypertension.
* Human immunodeficiency virus (HIV) positivity.
* Active hepatitis (hep) B or C or other active liver disease.
* Persistent clinically significant toxicity from prior chemotherapy that is Grade 2 or higher by the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE v3) (see Inclusion Criteria).
* Drugs (or medical conditions) that are generally accepted to have a risk of causing torsades de pointes (see Appendix E). Subjects who have discontinued any of these medications must have a wash-out period of at least 5 days or 5 half-lives of the drug (whichever is greater) prior to the first dose of AC480.
* Proton pump inhibitors and histamine H2 antagonists. Other antacid agents may be taken, but not within 8 hours before or 4 hours after dosing of AC480. A detailed log recording administration of other antacids in relation to AC480 must be kept.
* Medical condition, serious intercurrent illness, or other extenuating circumstance that, in the judgment of the Principal Investigator, could jeopardize subject safety or interfere with the objectives of the study.
* Patient is < 3 years free of another primary malignancy except: if the other primary malignancy is not currently clinically significant or requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ.
* Concurrent administration of warfarin, rifampin or St. John's Wort, except for low-dose warfarin (1mg po DAILY).
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-11; Primary Completion 2010-10 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Intratumoral and plasma pharmacokinetics of AC480 will be obtained on surgical tissue specimens from 5 patients treated pre-operatively with AC480. | At time of resection

SECONDARY OUTCOMES:
Anti-proliferative effect of AC480 by FDG-PET | 2 weeks
Intratumoral and plasma pharmacodynamics of AC480 | 6 months
6-month progression-free survival (PFS) | 6 months
Radiographic response | 6 months
Adverse event and toxicity monitoring | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, FRCPC, Principal Investigator — Duke Health
Locations (1):
- The Preston Robert Tisch Brain Tumor Center at Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center — http://www.cancer.duke.edu/btc/